CLINICAL TRIAL: NCT06787768
Title: User Experience of a Technology Based Rehabilitation Programme
Brief Title: Technology Enriched Rehabilitation Gym
Acronym: TERG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Strathclyde (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UStrathclyde_UEC20/08 Kerr
Record Dates: First submitted 2024-08-14; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Stroke; Rehabilitation
Keywords: Rehabilitation; Technology
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Two baselines measures of function (mobility) separated by 14 days recorded at least 1 week before the intervention. Intervention is an 8 week rehabilitation programme delivered with technology. Measures of function repeated immediately after intervention
Masking Description: No masking is used
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Chronic stroke survivors (Experimental): People well enough to exercise lightly but living with motor impairment following a stroke at least 12 months previously
  Interventions: Other: Technology Enriched Rehabilitation Gym

INTERVENTIONS:
Other: Technology Enriched Rehabilitation Gym — The intervention is an 8-week long rehabilitation programme delivered entirely through technology, including virtual reality (immersed and non-immersed), treadmills, weight suspension and movement resistance, and power assistance equipment located in a gym-like space on a university campus. Individual programs are designed, supervised, and reviewed by a physiotherapist using principles of intensity, feedback, cognitive engagement, and aerobic activity to address the goals identified by the participant and scores from outcome measures at baseline. Participants attend a minimum of two times per week and can attend daily for the two hour group based circuit class.

SUMMARY:
The department (Biomedical Engineering, University of Strathclyde) co-creates rehabilitation technology. To improve the quality of the feedback the investigators have set up a programme of rehabilitation supervised by qualified therapists (physical therapists, occupational therapists and speech therapists) and delivered entirely through technology. This tests the feasibility of the overall approach as well as helping develop specific pieces of equipment.

DETAILED DESCRIPTION:
A key area of research activity within the Biomedical Engineering Dept. is the development of rehabilitation technologies to support the recovery of function in people with movement disorders such as stroke, cerebral palsy and spinal chord injury. A critical part of the design process for these technologies is the close involvement of users from concept through to prototype testing. Despite significant levels of investment rehabilitation technologies continue to experience barriers to adoption among private users and the health service with issues such as cost, usability, portability and accessibility cited as factors. Adopting a partnership approach towards the development of these technologies would address these issues.

Engagement between technology designers and users is typically ad-hoc and project specific with users invited to attend design concept workshops or "try out" sessions with a technology in the prototype stages of its development. While these experiences are certainly useful they are unable to provide the in-depth information needed to inform the translation of these technologies into practice, neither do they provide the interactions capable of generating new ideas.

The aim of this project is to test the feasibility of a technology enriched rehabilitation programme in people living with stroke and gather user feedback on specific technology. The programme offers professionally supervised (therapists) access to an existing suite of commercially available and prototype rehabilitation technologies for 8 weeks, 2-5 times a week. Such an arrangement provides a critical source of feedback as well as creating considerable opportunity for new ideas to emerge, both for specific technologies and models of delivery. Specifically it would:

1. Provide stroke survivors with time limited, professionally supervised, access to an integrated suite of rehabilitation technologies.
2. Enable data to be collected from users on their response to the intervention. This would include:

   * Demographics (age, gender)
   * Stroke detail (number of strokes and time since last stroke).
   * Stroke related impairments in mobility, speech and cognition
   * Co-morbidities (number and nature).
   * Change in impairments as a response to the rehabilitation intervention
3. Collect data on their interactions and general experiences with the rehabilitation technologies.

This would include a recorded interview at the end of their participation covering opinions on specific technologies and general views on the use of technology in the rehabilitation process including access. It will also conduct focus groups (n=5 to 8) to explore the use of goal setting and the development of an educational package to help individuals continue their rehabilitation after the programme completes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stroke at least 12 months previously
* Currently well
* Not currently receiving rehabilitation
* Able to attend the programme for two hours at least twice a week
* Able to follow instructions in English and follow provide verbal and/or written feedback

Exclusion Criteria:

* Absolute contradictions to physical activity
* Recent (6 weeks) deterioration in health
* Change in medication
* Currently unwell

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
10-meter walk test (10mWT) | Four time points; 1) Two weeks before intervention starts,2) immediately before the intervention, 3) week 4 (halfway way through intervention) and 4) immediately after intervention ends
  Time to walk 10 metres

CONTACTS AND LOCATIONS:
Overall Officials: Milena Sklachetka, BSc, Principal Investigator — University of Strathclyde
Locations (1):
- University of Strathclyde, Glasgow, Glasgow, United Kingdom